CLINICAL TRIAL: NCT03440073
Title: Mulligan Concept Intervention for Pregnancy Related Lumbo Pelvic Pain
Brief Title: Intervention for Pregnancy Related Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Idaho (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-042; 18-22QR-UI-PG76 (Other Grant/Funding Number: Clinical Translational Research Infrastructure Network)
Record Dates: First submitted 2018-02-01; First posted 2018-02-20 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Other Specified Pregnancy-Related Conditions
Keywords: pregnancy; pain; pelvis; spine; manual therapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Concept Intervention (Experimental): Mulligan Concept Intervention, including Mobilizations with Movement intervention is administered. Up to 30 minutes total treatment time.
  Interventions: Other: Mulligan Concept Intervention
- Sham Mulligan Concept Treatment (Sham Comparator): Assessment procedures of the Mulligan Concept are followed, but no manual pressure is applied to the participant during treatment to provide a sham Mulligan Concept Treatment.
  Interventions: Other: Sham Mulligan Concept Treatment

INTERVENTIONS:
Other: Mulligan Concept Intervention — The concept is a manual therapy paradigm that includes a clinician applying joint mobilizations and having the patient perform concurrent active, pain free, movement.
  Arms: Mulligan Concept Intervention
Other: Sham Mulligan Concept Treatment — The treating clinician will ask the participant to perform the movements associated with the Mulligan Concept technique. The clinician will have her hands on the participant during the movement but will not apply any pressure or force.
  Arms: Sham Mulligan Concept Treatment

SUMMARY:
Women in rural communities receive less access to prenatal care, and experience slightly higher rates of complications during pregnancy. A very prevalent pregnancy related complication is Pregnancy Related Pelvic Girdle Pain (PPGP), effecting up to 76% of all pregnant women. Historically, PPGP has been thought to originate from hormonal changes associated with pregnancy, but its cause is more likely due to loss of motor control and/or malpositioning of the pelvic bones. Despite growing interest and clinical awareness of the condition, treatment outcomes of PPGP are inconsistent and intervention studies are lacking. The goal of this proposal is to investigate a treatment modality with minimal risks and potential to be self-administered. The Mulligan Concept manual therapy technique aims to restore mechanical function of the lumbopelvic region and has yet to be measured in women with PPGP.

DETAILED DESCRIPTION:
The long-term goal of this project is to develop an effective conservative treatment protocol that is easily accessible. The objective of this application is to determine if patients who are treated with Mulligan Concept manual therapy experience immediate and significant changes in pain and function. Our specific aims are: In women with PPGP, 1.) Determine if Mulligan Concept treatment produces immediate changes in pain and function, 2.) Determine whether the Mulligan Concept immediately restores or alters dysfunctional gait characteristics and pelvic girdle motor control, and 3.) Identify factors that mathematically predict treatment outcome. Our central hypothesis is that restoration of lumbopelvic positioning will result in immediate decrease in pain, increase in function, and improved gait mechanics.

Volunteers in the 20th-34th week of pregnancy, ages 20-45 years, who are experiencing PPGP will be screened and randomly assigned into treatment or placebo group based on age, weight, height, gestational week and number of pregnancies. All participants will undergo a standardized examination, complete patient reported outcome measures, and perform a walking gait, sit to stand, and active straight leg raise tasks. Kinematic, kinetic, and EMG recordings will be taken during performance of the tasks. The participants of the treatment group will receive a Mulligan Concept evaluation and treatment. Participants in the placebo group will receive only the Mulligan Concept evaluation. Participants will then repeat the same tasks and measures. The study will be conducted under a randomized triple blinded placebo trial design; the patients, researchers, and treating clinician will be blinded to group assignment. Independent sample t-tests will be conducted to determine if significant differences exist between the intervention and placebo group across several dependent variables. Regression analysis will be conducted in order to determine if intake factors mathematically predict treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* reported pregnancy-related lumbopelvic pain

Exclusion Criteria:

* orthopaedic or neurological problems with walking
* prior surgery of the lumbar spine, pelvis, hip, or knee
* fracture
* known malignancy
* active inflammation in the lumbar spine or pelvis
* ankylosing spondylitis, Scheuermann's kyphosis, active polyarthritis, or severe osteoporosis
* any pulmonary, cardiac, visual, auditory, or cognitive disorders
* any other multi/co-morbidities that limit the volunteers ability to complete a gait and sit-to-stand task
* does not receive consent from their maternity care provider
* pain is associated with something other than pregnancy, or is experienced outside of pregnancy prior to the first pregnancy

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
3-D motion Analysis- sit to stand | Change from pre to post intervention (immediate, 30 minutes)
  Kinematic data is collected during sit to stand task
3-D Motion Analysis- gait | Change from pre to post intervention (immediate, 30 minutes)
  Kinematic data is collected during gait task
3-D Motion Analysis- active straight leg raise | Change from pre to post intervention (immediate, 30 minutes)
  Kinematic data is collected during active straight leg raise task

SECONDARY OUTCOMES:
Electromyography- Sit to Stand | Change from pre and post intervention (Immediate, 30 minutes)
  EMG data will be collected during the sit to stand task
Electromyography- Gait | Change from pre and post intervention (Immediate, 30 minutes)
  EMG data will be collected during gait task
Electromyography- Straight Leg Raise | Change from pre and post intervention (Immediate, 30 minutes)
  EMG data will be collected during the sit to stand, gait, and active single leg raise tasks.
Visual Analog Pain Scale | Change from pre and post intervention (Immediate, 30 minutes)
  Patient Reported Outcome Measure, pain
Pelvic Girdle Questionnaire | Change from pre and post intervention (Immediate, 30 minutes)
  Patient Reported Outcome Measure, region specific disablement
Assessment of Disablement Questionnaire | Change from pre and post intervention (Immediate, 30 minutes)
  Patient Reported Outcome Measure, global disablement
Short Stress State Questionnaire | Change from pre and post intervention (Immediate, 30 minutes)
  Patient Reported Outcome Measure, stress

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Larkins, DAT, Principal Investigator — University of Idaho
Locations (1):
- Integrated Sport Medicine and Rehabilitative Therapy Clinic, Moscow, Idaho, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be known to the PI. Other researchers working on the project are blinded to IPD. The PI will maintain records on a secure computer, with secure server connection, located in a locked office. Data will be shared in aggregate without identifying information.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03440073/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03440073/ICF_001.pdf